CLINICAL TRIAL: NCT01725776
Title: Pharmacokinetic and Pharmacodynamic of Inhaled Milrinone in Cardiac Surgical Patients
Brief Title: Inhaled Milrinone in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government); St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Andre Denault, MD PhD FRCPC ABIM-CCM, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM 06-888
Record Dates: First submitted 2012-06-18; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Cardiac surgery; Cardiopulmonary Bypass (CPB)
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Milrinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhaled milrinone 5 mg (Experimental): Inhaled milrinone 5 mg(as for the injectable solution)
  Interventions: Drug: Inhaled milrinone 5 mg

INTERVENTIONS:
Drug: Inhaled milrinone 5 mg — Inhaled milrinone 5 mg (as for the injectable solution)
  Other Names: Primacor

SUMMARY:
The purpose of this study is to investigate the concentration-effect relationship of inhaled milrinone after prophylactic administration in cardiac surgical patients with preoperative pulmonary hypertension undergoing cardiopulmonary bypass.

DETAILED DESCRIPTION:
Milrinone elimination will be verify with blood and urine samples analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac surgery under CPB
* High risk patients: NYHA class II-III
* Preoperative diagnostic of pulmonary hypertension:

  * Systolic pulmonary artery pressure (sPAP) > 35 mm Hg; or
  * Mean pulmonary artery pressure (mPAP) > 25 mm Hg; or
  * mAP/mPAP < 3.0 (after induction of anesthesia).

Exclusion Criteria:

* Open Heart Surgery
* Contraindication to transesophageal echocardiography (TEE)
* Hemodynamic instability before surgery
* Emergency surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Study the elimination rate of milrinone administered by inhalation | up to 24 hours

SECONDARY OUTCOMES:
Demonstrate the presence or absence of hemodynamic and echographic effects observed after inhalation of milrinone | 15 min after the of study drug administration
  hemodynamic values evaluated will be: central venous pressure, systolic and diastolic pulmonary pressure, wedge, cardiac output, cardiac frequency, systolic and diastolic pressure, SaO2, EtCO2. Patient will also have arterial and venous gaz. Echographic values will be evaluated to see the cardiac fonction: left and right ventricular systolic and diastolic function and valvular function.
Confirmation of the safety of inhaled milrinone | 24 hours after cardiac surgery
  Verification of the absence of deleterious effects on cardiac output and systemic arterial pressure.
Determination of the efficacy of inhaled milrinone in the treatment of pulmonary hypertension | 15 min after end of milrinone administration
  Efficacy in the treatment of pulmonary hypertension is defined as a reduction of the mean pulmonary pressure of 10-20 %

CONTACTS AND LOCATIONS:
Overall Officials: Andrée Denault, MD PhD FRCPC, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada